CLINICAL TRIAL: NCT06192732
Title: Environmentally Sustainable Nutrition for Older Adults (55+) With Obesity: a Pilot Study
Brief Title: Environmentally Sustainable Nutrition for Older Adults (55+) With Obesity
Acronym: 2EAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amsterdam University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAAK.PRO04.033
Record Dates: First submitted 2023-12-12; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Obesity; Aging
Keywords: Obesity; Older adults; Healthy ageing; Sustainability; Plant-based protein; Plant-based diet; Sustainable diets; Dietary counseling
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- More plant-based diet (Experimental): Participants receive the dietary counselling focused on a more plant-based diet during weight loss
  Interventions: Behavioral: A more plant-based diet during weight loss

INTERVENTIONS:
Behavioral: A more plant-based diet during weight loss — Participants receive dietary counseling on a more plant-based diet during weight loss. They will be counseled by a dietician to increase their plant-based protein intake up to 60%, focusing on 1.2 grams of protein per kg body weight.

SUMMARY:
The objective of the pilot study (feasibility study) is to assess the acceptability and feasibility of the developed 2EAT dietary treatment in obese older adults (55+).

For ecological reasons, the goal of the dietary treatment plan is to achieve an intake of 60% plant-based proteins in older adults (55+) in a healthy and nutritionally adequate way during a period of weight loss. The investigators developed the new dietary treatment plan for 6 months (RCT). To further optimize the new treatment plan the 2EAT study includes this feasibility study with a duration of 8 weeks.

In the feasibility study, the effect of a more plant-based hypocaloric diet on the protein intake of older adults (55+) with obesity is evaluated. To assess the feasibility of the treatment plan, 20 obese older adults will follow the newly developed dietary treatment for 8 weeks. The participants will be guided by experienced dieticians that are part of the study consortium, in their dietetic practice. All dieticians will be trained to execute the 2EAT dietary treatment plan.

The desired effect of the treatment is that participants change their protein intake and achieve an intake of 1.2 g/kg/d of which 60% is from plant-based sources. Additionally, the experience of both the older adults as well as the experience of the dieticians will be monitored during the 8 weeks of intervention. During 8 weeks there will be continuous monitoring of the implementation of the treatment plan by keeping logbooks (dieticians), and measurement of the food intake of the participants. When participants deviate from the diet, the dietician must make timely adjustments with available behavioral techniques. The primary outcome of the feasibility phase is the protein intake: source (plant-based vs. animal-based), amount (g/kg/day) and protein quality per meal (amino acid score). Secondary outcomes are the body weight and BMI of participants and qualitative information about the experience of participants and dieticians with the use of the new treatment plan. Dieticians are professionals in working with older clients with obesity during a weight loss program, and are competent to execute the treatment plan and additionally monitor and make adjustments to coach the participant towards the desired diet and goal. Findings and experiences from the 8-week feasibility study will be used to further improve the 2EAT dietary treatment. The optimized dietary plan will eventually be used in the RCT study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 or older
* Are obese: have a BMI of >30 kg/m2 or BMI >27 kg/m2 and waist circumference >88 cm (women) or >102 cm (men)
* Living independently (not in a health facility)
* The willingness that the general practitioner will be notified of study participation
* Written informed consent
* Willingness to comply with the protocol
* Consent of the study physician

Exclusion Criteria:

* Inability to understand the Dutch language
* Cognitive impairment (MMSE <15)
* Use of total or partial parenteral nutrition (TPN)
* Alcohol or drug abuse in the opinion of the investigator
* Current enrolment in a fixed rehabilitation program or other intervention studies
* Palliative treatment or a life expectancy of ≤ 3 months
* Following a vegan (100% plant-based) diet
* Active medical treatment interfering with this intervention (e.g. cancer patients receiving systemic and immune therapy)
* Physical disabled: unable to meet the general daily exercise guideline for adults
* Planned a holiday during the intervention period and is unable to attend group- or individual sessions for > 1 week

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility | Baseline (week 0) and endline (week 9)
  The objective of the feasibility study is to assess the feasibility of the developed 2EAT dietary treatment in obese older adults (55+). The feasibility focusses on the ratio plant-based and animal-based protein, where it is aimed to reach 60% plant-based proteins at endline (week 9). This will be investigated via 3-day dietary records (measured at baseline and endline).
Assess the acceptability | Endline (week 9)
  The objective of the feasibility study is to assess the acceptability of the developed 2EAT dietary treatment in obese older adults (55+). This will be investigated via focus groups. Focus groups will be organized for participants and dieticians separately at endline (week 9).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Weijs, Principal Investigator — Amsterdam University of Applied Sciences

IPD SHARING:
Plan to Share IPD: No